CLINICAL TRIAL: NCT04970992
Title: A Pharmacokinetic and Pharmacodynamic Study of DZ-002 in Patients With Advanced Solid Malignancies or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Da Zen Theranostics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DZ-002-101
Record Dates: First submitted 2021-07-07; First posted 2021-07-21 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Solid Tumor; Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose escalation and cohort expansion Q1W (Experimental): DZ-002 treatment once every week
  Interventions: Drug: DZ-002

INTERVENTIONS:
Drug: DZ-002 — DZ-002 Injection

SUMMARY:
The primary goal of this Phase 1 study is to characterize the safety and tolerability of DZ-002 and establish the maximum tolerated dose (MTD) and the recommended Phase 2 dose (RP2D) of DZ-002 administered on a weekly schedule in patients with solid tumors. Pharmacokinetics, pharmacodynamics, and the anti-tumor activity of DZ-002 will also be assessed.

DETAILED DESCRIPTION:
This is a single center, first-in-human, Phase 1, safety, PK and pharmacodynamic study of DZ-002 in patients with solid tumors who have failed standard therapies. The study will be conducted in 2 phases, a dose escalation phase and a dose expansion phase. The dose-escalation phase will first determine the MTD and/or RP2D of DZ-002 in patients with advanced cancers. Subsequently, the MTD and/or RP2D will be investigated in 2 expansion treatment groups of castration-resistant prostate cancer (CRPC) and advanced pancreatic cancer. Patients who are determined to be eligible, based on Screening assessments, will be enrolled in the study and will receive their first dose of study therapy on Cycle 1 Day 1. All patients will receive DZ-102 administered as a weekly intravenous (IV) infusion on days 1, 8, 15, and 22 of a 28-day cycle. The dose of DZ-002 will be dependent on the cohort in which the patient is enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically confirmed diagnosis of an advanced, unresectable, or metastatic solid malignant tumor (including lymphoma; dose-escalation phase only) that has failed to respond to standard therapies;
2. Male or female patients age 18 or older;
3. Measurable or evaluable disease by RECIST v 1.1, or PCWG3 for prostate cancer;
4. Capable of understanding and complying with protocol requirements;
5. A life expectancy of greater than 8 weeks at Screening;
6. An ECOG PS of 0 to 2;
7. Written informed consent from the patient or the patient's legally acceptable representative prior to the initiation of any study procedures;
8. Adequate bone marrow, liver, and renal function as defined below:

   * Hemoglobin ≥ 8.0 g/dL (transfusions and/or erythropoietic stimulating growth factors allowed);
   * Absolute neutrophil count ≥ 1500/μL;
   * Platelet count ≥ 75,000/ μL;;
   * Alanine aminotransferase and aspartate aminotransferase ≤ 2.5 × the upper limit of normal (ULN) or ≤ 5 × ULN for patients with known hepatic metastases;
   * Total serum bilirubin ≤ 1.5× ULN or ≤ 2 .0 × ULN if liver metastases are present. Patients with a known history of Gilbert's syndrome (≤ 3.0 × ULN) and/or isolated elevations of indirect bilirubin are eligible for study participation;
   * Estimated creatinine clearance ≥ 40 mL/min(using the Cockcroft Gault formula);
9. Adequate cardiac function as estimated by left ventricular ejection fraction (LVEF) > 50% by multiple-gated acquisition (MUGA) or echocardiogram (ECHO);
10. Negative pregnancy test for women of childbearing potential (women of childbearing potential and men must agree to use adequate contraception [hormonal or barrier method of birth control] prior to study entry and for the duration of study participation.

[NOTE: Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study intervention. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the patient]. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately).

Exclusion Criteria:

1. New York Heart Association (see Appendix 5) Class III or IV cardiac disease, myocardial infarction within the past 6 months, unstable arrhythmia, a history of risk factors for Torsades de Pointes, including heart failure, hypokalemia, and family history of long QTc syndrome, or evidence of ischemia on ECG;
2. Baseline QTc exceeding 470 msec (using the Fridericia's formula) and/or patients receiving Class 1A or Class III antiarrhythmic agents or concomitant medications that prolong the QT/QTc interval;
3. Active, uncontrolled bacterial, viral, or fungal infections requiring systemic therapy;
4. Treatment with simvastatin unless it can be stopped prior to and during the study.
5. Treatment with strong inhibitors and inducers of CYP3A4 or narrow therapeutic index substrates of CY3A4, CYP2B6, CYP1A2, CYP2C9 and CYP2C8, unless these can be stopped prior to and during the study
6. Known sensitivity to DZ-002 or drug excipients
7. Pregnant (confirmed by serum or urine pregnancy test) or is breast feeding;
8. Treatment with radiation therapy, surgery, chemotherapy, or investigational therapy within 30 days prior to study entry (6 weeks for nitrosoureas or Mitomycin C);
9. Unwillingness or inability to comply with procedures required in this protocol;
10. Known infection with human immunodeficiency virus and CD4 lymphocyte count < 200 cells/mm3 , or active hepatitis B virus, or hepatitis C virus infections;
11. Serious nonmalignant disease (e.g., hydronephrosis, liver failure, or other conditions) that could compromise protocol objectives in the opinion of the investigator and/or the Sponsor;
12. Patients who are currently receiving any other investigational agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment emergent adverse events (TEAEs) | 24 months
  Safety is based on evaluation of adverse events (AEs) and serious adverse events (SAEs) from the time of study drug administration through the End of Study visit
MTD | 24 months
  maximum tolerated dose (MTD) of DZ-002

SECONDARY OUTCOMES:
Tumor response | 24 months
  Tumor response as defined by Response Evaluation Criteria in Solid Tumors (RECIST v1.1) and the Prostate Cancer Working Group 3 (PCWG3) for prostate cancer
AUC | 56 days
  Area Under the Plasma Concentration versus Time Curve of DZ-002
Cmax | 56 days
  Maximum Plasma Concentration of DZ-002
Tmax | 56 days
  Time to reach maximum (peak) plasma concentration of
t1/2 | 56 days
  Terminal half-life of DZ-002
Clearance | 56 days
  Total body clearance of the drug from plasma (CL) of DZ-002
Volume of distribution | 56 days
  Apparent volume of distribution of DZ-002

CONTACTS AND LOCATIONS:
Overall Officials: Robert L De Jager, MD, Study Director — Dazen Theranostics
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States